CLINICAL TRIAL: NCT04037683
Title: An Alongside Qualitative Study Exploring Patients' and Health Care Professionals' Expectations and Experiences of Labour Induction With Misoprostol and Oxytocin for Hypertension in Pregnancy in India
Brief Title: qMOLI- A Qualitative Assessment of Misoprostol or Oxytocin for Labour Induction
Acronym: qMOLI
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Government Medical College, Nagpur (Industry); Gynuity Health Projects (Other)
Responsible Party: Principal Investigator, Andrew D Weeks, Professor of International Maternal Health, University of Liverpool
Other Study IDs: 4791
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Pre-Eclampsia
Keywords: induction of labour; intrapartum fetal monitoring; qualitative; semi-structured interview; focus groups
MeSH Terms: conditions — Pre-Eclampsia | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MOLI participants pre IOL: Semi-structured interviews with MOLI participants - estimated 12 patients (until data saturation) after recruitment to MOLI RCT but prior to the start of the induction of labour (IOL) process
- MOLI participants post IOL (misoprostol/misoprostol): Semi-structured interviews with MOLI participants - estimated 12 patients (until data saturation) 12 women post IOL with misoprostol/misoprostol Semi-structured interviews with MOLI participants - estimated 12 patients (until data saturation) 12 women post IOL with misoprostol/oxytocin
  Interventions: Drug: Misoprostol Oral Tablet
- MOLI participants post IOL (misoprostol/oxytocin): Semi-structured interviews with MOLI participants - estimated 12 patients (until data saturation) 12 women post IOL with misoprostol/oxytocin
  Interventions: Drug: Misoprostol Oral Tablet; Drug: Oxytocin
- Staff focus group pre and during MOLI recruitment: A focus group in each of the 2 recruitment sites before the start of the MOLI trial (n=2) A focus group in each of the 2 recruitment sites and with each cadre of staff during the MOLI trial (n=8)
  * Research assistants
  * Residents
  * Consultants
  * Midwives

INTERVENTIONS:
Drug: Misoprostol Oral Tablet — Misoprostol 25mcg orally given 2-hourly
  Groups: MOLI participants post IOL (misoprostol/misoprostol); MOLI participants post IOL (misoprostol/oxytocin)
Drug: Oxytocin — Oxytocin infusion
  Groups: MOLI participants post IOL (misoprostol/oxytocin)

SUMMARY:
Q MOLI is an alongside qualitative study, for the 'Misoprostol or Oxytocin for Labour Induction' (MOLI) pragmatic, open-label, randomised controlled trial, comparing a misoprostol/misoprostol regime vs the standard misoprostol/oxytocin induction of labour regime.1000 patients with hypertensive disease in pregnancy will be recruited, over 24 months, in Nagpur, India.

DETAILED DESCRIPTION:
Qualitative study involving semi-structured interviews, with participants (pregnant women with hypertension/pre-eclampsia participating in the 'Misoprostol or Oxytocin for Labour Induction' (MOLI) study who consent to enter the qualitative study) in a randomised trial, pre and post induction of labour and focus group discussions with healthcare professionals involved in the study (MOLI study staff; practitioners who are involved in screening, recruiting, randomising and consenting participants to the MOLI study).

The investigators aim to assess the priorities, experiences and acceptability of women being induced for hypertension in pregnancy in India, and clinician's views on the feasibility, usability, acceptability and barriers to implementation of various induction protocols.

1. Explore patients' perceptions, expectations, priorities, understanding of and concerns around induction of labour, prior to induction.
2. To explore the experiences, acceptability and satisfaction of patients post induction and any differences between the two RCT groups; misoprostol/misoprostol vs misoprostol/oxytocin regimes.
3. To better understand the feasibility, usability and acceptability of the different induction regimes to health care professionals. To explore potential barriers for implementing research findings into clinical practice and potential solutions.
4. To explore patients' and staff perspectives of the fetal monitoring regimens during the induction process.

ELIGIBILITY:
MOLI RCT participants (women being induced)

Inclusion criteria

* Women who are recruited to the MOLI RCT and are either antenatal, or post-induction and meet all of the eligibility criteria:
* Women who consent to join the qualitative study

Exclusion criteria

* Women who are not recruited to the MOLI RCT
* Women who lack the capacity to make an informed decision
* Women under the age of 16
* Women who have had a stillbirth in this pregnancy
* Women who are distressed/in pain
* Women too unwell to take part in interviews, or who need urgent intervention (in less than 2 hours)
* Where delay in starting the IOL process due to time of interview could cause harm to the patient
* Women who do not give consent to be in the study

MOLI practitioners

Inclusion criteria

• Practitioners who are involved in screening, recruiting, randomising and consenting participants to MOLI RCT

Exclusion criteria

* Staff who do not wish to be included
* Staff who do not give their consent to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant or postnatal women with hypertension/pre-eclampsia participating in the 'Misoprostol or Oxytocin for Labour Induction' (MOLI) study who consent to enter the qualitative study.
  MOLI study staff. Practitioners who are involved in screening, recruiting, randomising and consenting participants to the MOLI study.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patients' views on induction of labour, prior to induction. | 6 months
  Explore patients' perceptions of induction of labour, prior to induction.
Patients' views on induction of labour, post induction. | 6 months
  To explore the experiences of patients post induction and any differences between the two RCT groups; misoprostol/misoprostol vs misoprostol/oxytocin regimes.
Clinicians' views on various induction protocols. | 6 months
  To better understand the acceptability of the different induction regimes to health care professionals. To explore potential barriers for implementing research findings into clinical practice and potential solutions.
Patients' views on the fetal monitoring regimens during the induction process. | 6 months
  To explore patients' perspectives of the fetal monitoring regimens during the induction process.
Staff's views on the fetal monitoring regimens during the induction process. | 6 months
  To explore staff perspectives of the fetal monitoring regimens during the induction process.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Weeks, Professor, Principal Investigator — University of Liverpool; Kate Lightly, Dr, Study Director — University of Liverpool
Locations (1):
- Government Medical College, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lightly K, Mundle S, Tripathy J, Deshmukh P, Winikoff B, Weeks A, Kingdon C. Women and clinicians' views, preferences and experiences of caesarean section and vaginal birth in India: a qualitative substudy of the 'Misoprostol or Oxytocin for Labour Induction' (MOLI) trial. BMJ Glob Health. 2025 Sep 5;10(9):e018393. doi: 10.1136/bmjgh-2024-018393. PMID 40912733